CLINICAL TRIAL: NCT00629837
Title: A Randomized, Double-blind, Cross-over Study to Determine the Pharmacokinetics and Safety of a Single Intravenous Infusion of BAY 79-4980 in Previously Treated Patients With Severe Hemophilia A
Brief Title: Pharmacokinetics and Safety of a Single Intravenous Infusion of BAY 79-4980
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11876; LipLong
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Hemophilia A
Keywords: FVIII; Long acting; pk
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Biological: Recomb. Factor VIII (Kogenate FS Liposome, BAY79-4980)
- Arm 2 (Experimental)
  Interventions: Biological: Recomb. Factor VIII (Kogenate FS Liposome, BAY79-4980)
- Arm 3 (Active Comparator)
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Arm 4 (Active Comparator)
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recomb. Factor VIII (Kogenate FS Liposome, BAY79-4980) — Low dose of BAY 79-4980 [13mg of liposomes/kg] then cross over to rFVIII-FS (35 IU/kg reconstituted in 2.5 mL WFI / 1000 IU).
  Arms: Arm 1
Biological: Recomb. Factor VIII (Kogenate FS Liposome, BAY79-4980) — High dose of BAY 79-4980 [22mg of liposomes/kg] then cross over to rFVIII-FS (35 IU/kg reconstituted in 2.5 mL WFI / 1000 IU)
  Arms: Arm 2
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — rFVIII-FS (35 IU/kg reconstituted in 2.5mL WFI /1000 IU) then cross over to low dose of BAY 79-4980 [13mg of liposomes/kg]
  Arms: Arm 3
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — rFVIII-FS (35 IU/kg reconstituted in 2.5mL WFI /1000 IU) then cross over to high dose of BAY 79-4980 [22mg of liposomes/kg]
  Arms: Arm 4

SUMMARY:
The primary objective of this study is to determine the pharmacokinetic profile after single administration of two doses of BAY 79-4980 (high and low: 35 IU FVIII/Kg reconstituted in 22 mg and 13 mg of liposomes/Kg, respectively) compared to rFVIII-FS (35 IU/Kg reconstituted in 2.5 mL WFI/1000 IU) in PTPs aged 12 to 60 years with severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 12 to 60 years
* Hemophilia A with plasma FVIII level less than 1% (severe hemophilia)
* No history of FVIII inhibitor antibody formation and no current evidence of inhibitor antibody measured using the Nijmegen modified Bethesda assay (< 0.6 Nijmegen Bethesda Units [N.B.U.]/mL)
* No signs or symptoms of an acute bleeding episode on the day of infusion
* Four or more days without treatment with FVIII prior to the day of infusion
* Subject (or the subject's legal representative) must provide written informed consent and authorization of use and disclosure of Protected Health Information (PHI)
* Subjects must have been previously treated with FVIII concentrate for a total of at least 200 exposure days, including 20 exposure days in the previous 12 months. Previous treatment can have been with any type of rFVIII or plasma-derived FVIII concentrate

Exclusion Criteria:

* Individuals with abnormal renal function (serum creatinine concentrations greater than 1.3 mg/dL) or active hepatic disease (persistent aspartate aminotransferase [AST] or alanine aminotransferase [ALT] increases to greater than five times the upper limit of normal).
* Individuals with anemia, as defined by hemoglobin level less than 12 g/dL
* Any individual with a past history of severe reaction(s) to FVIII products
* Any individual on interferon treatment or who has received interferon within the previous 3 months
* Any individual with thrombocytopenia (platelets greater than or equal to 100,000 cells/mm3) or known hematologic/bleeding problems other than hemophilia A
* Any individual who is receiving or has received other experimental drugs within 3 months prior to study entry
* Any individual with known dislipidemic disease or actively taking cholesterol lowering drugs for the treatment of hypercholesterolemia or hyperlipidemia (e.g., statins, cholesterol absorption inhibitors, bile acid sequestrants, nicotinic acid or fibrates) or individuals taking anaesthetic drugs
* Any individual who requires pre-medication for FVIII infusions (e.g., antihistamines)
* Any individual with high blood pressure (defined as diastolic blood pressure great than or equal to 100 mm/Hg)
* Any patient who cannot forego FVIII treatment for at least 4 days prior to study entry or between study infusions due to a need for more frequent prophylactic treatment because of a pre-existing medical condition
* Any patient with known allergy or severe reactions to liposomes or PEG
* Individuals with any other known disease affecting hemostasis besides hemophilia A
* Any patient who is not suitable for participation in this trial for any reason, according to the Investigator

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2005-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the pk profile after single administration of two doses of BAY 79-4980 (high and low: 35 IU FVIII/Kg reconstituted in 22 mg and 13 mg of liposomes/kg, respectively) compared to rFVIII-FS (35 IU/Kg reconstituted in 2.5 mL WFI/1000 IU) in PTPs | 6 weeks

SECONDARY OUTCOMES:
To determine the infusion tolerability of both BAY 79-4980 doses, by evaluation of vital signs and adverse events | 6 weeks
To determine the safety of both BAY 79-4980 doses by measuring the effects on laboratory parameters - especially the lipid profile and adverse events | 6 weeks
To determine the pk characteristics of liposomes - esp body clearance by measuring the major liposome component 1-palmitoyl-2-oleoyl-sn-glycerol-3-phosphocholine (POPC) and the non-biological liposome component, MPEG 2000 DSPE, as surrogate marker | 6 weeks
To determine the activity of rFVIII over time (as determined by thrombin generation assay and the rotation thromboelastography [RoTEG] assay) for both doses of BAY 79-4980 compared to rFVIII-FS | 6 weeks
Additional analyses of the number and timing of spontaneous bleeds after each study treatment will be assessed | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Davis, California
  - Orange, California